CLINICAL TRIAL: NCT04797858
Title: Secondary Distribution of COVID-19 Self-tests vs. Referrals to Increase Test Uptake in Underserved Populations
Brief Title: COVID-19 Self-Testing Through Rapid Network Distribution
Acronym: C-STRAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Public Health Management Corporation (Other)
Responsible Party: Principal Investigator, Robert Gross, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 3R01HL151292-01S1 (NIH)
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Test kit distribution (Experimental): Participants in the self-test arm receive multiple COVID-19 self-test kits to distribute to others in their social networks.
  Interventions: Behavioral: COVID-19 self-test
- Test referral distribution (Active Comparator): Participants in the test referral arm receive multiple COVID-19 test referral cards and text messages to distribute to others in their social networks.
  Interventions: Behavioral: COVID-19 test referral

INTERVENTIONS:
Behavioral: COVID-19 self-test — 5 COVID-19 self-test kits will be given to participants after they have been tested for COVID-19. Participants will be instructed to give test kits to others in their social networks who are symptomatic, exposed to COVID-19, or otherwise at high risk of COVID-19.
  Arms: Self-Test kit distribution
Behavioral: COVID-19 test referral — 5 test referral cards and text messages on how to obtain COVID-19 testing will be given to participants after they have been tested for COVID-19. These cards and text messages will have information on how to obtain free COVID-19 tests at local testing sites. Participants will be instructed to give out referral cards and text messages to others in their social networks to obtain testing.
  Arms: Test referral distribution

SUMMARY:
COVID-19, the coronavirus disease caused by SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2), has led to a global pandemic and has exacerbated existing health inequities among vulnerable populations. Despite higher rates of COVID-19 in Black and Latinx individuals compared to White individuals, rates of testing in predominately non-White, low-income communities are significantly lower than in high-income areas. Self-testing, where individuals collect their own samples, is now feasible for the detection of SARS-CoV-2. One promising approach to increase test uptake is the secondary distribution of self-testing kits, where an individual distributes tests to contacts in their social network and encourages them to self-test.

The central hypothesis of this clinical trial is that the secondary distribution of SARS-CoV-2 self-tests can significantly expand test uptake among underserved populations. To test this hypothesis, the investigators will conduct a 1:1 randomized controlled trial that will assess a self-testing intervention that promotes the secondary distribution of SARS-CoV-2 test kits compared with test referrals, with a focus on reaching underserved populations.

DETAILED DESCRIPTION:
Strategies to rapidly disseminate COVID-19 testing are urgently needed, particularly to address increasing health disparities among underserved communities. One promising approach to increase test uptake is the secondary distribution of self-tests, where an individual distributes test kits to contacts in their social network and encourages them to self-test. By decentralizing testing, this approach does not require individuals to have contact with medical systems, and can lower potential barriers to obtaining testing. This approach can increase case detection by facilitating testing among exposed individuals, and potentially ameliorate stigma, fear, and medical mistrust associated with COVID-19 among vulnerable populations because the testing process is decentralized.

The investigators will conduct a 1:1 randomized controlled trial randomizing individuals to receive either multiple self-test kits to distribute within their social circles, or referrals for standard clinic-based tests. All study participants will be offered testing upon enrollment. Study participants, deemed "Index Participants," will be randomized to receive multiple self-testing kits (intervention) or test referral cards and text messages (control) to encourage individuals in their social networks, deemed "network contacts" to test. Participants will complete a baseline evaluation and a follow-up evaluation at 8 weeks. We will measure network contact test uptake in both study arms. The central hypothesis of this trial is that distribution of self-test kits will increase test uptake compared with distribution of test referrals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has a working telephone number
* Willing and able to provide informed consent

Exclusion Criteria:

* Younger than 18 years of age
* Does not have a working telephone number
* Prior COVID-19 infection in the past 90 days
* Previously received a COVID-19 test as part of this COVID-19 research study
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gross, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Public Health Management Corporation, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bien-Gund C, Dugosh K, Acri T, Brady K, Thirumurthy H, Fishman J, Gross R. Factors Associated With US Public Motivation to Use and Distribute COVID-19 Self-tests. JAMA Netw Open. 2021 Jan 4;4(1):e2034001. doi: 10.1001/jamanetworkopen.2020.34001. PMID 33471114
- [Background] Lightfoot MA, Campbell CK, Moss N, Treves-Kagan S, Agnew E, Kang Dufour MS, Scott H, Sa'id AM, Lippman SA. Using a Social Network Strategy to Distribute HIV Self-Test Kits to African American and Latino MSM. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):38-45. doi: 10.1097/QAI.0000000000001726. PMID 29771792
- [Background] Golden MR, Kerani RP, Stenger M, Hughes JP, Aubin M, Malinski C, Holmes KK. Uptake and population-level impact of expedited partner therapy (EPT) on Chlamydia trachomatis and Neisseria gonorrhoeae: the Washington State community-level randomized trial of EPT. PLoS Med. 2015 Jan 15;12(1):e1001777. doi: 10.1371/journal.pmed.1001777. eCollection 2015 Jan. PMID 25590331
- [Background] Bagcchi S. Stigma during the COVID-19 pandemic. Lancet Infect Dis. 2020 Jul;20(7):782. doi: 10.1016/S1473-3099(20)30498-9. No abstract available. PMID 32592670
- [Background] MacGowan RJ, Chavez PR, Borkowf CB, Owen SM, Purcell DW, Mermin JH, Sullivan PS; eSTAMP Study Group. Effect of Internet-Distributed HIV Self-tests on HIV Diagnosis and Behavioral Outcomes in Men Who Have Sex With Men: A Randomized Clinical Trial. JAMA Intern Med. 2020 Jan 1;180(1):117-125. doi: 10.1001/jamainternmed.2019.5222. PMID 31738378
- [Background] Altamirano J, Govindarajan P, Blomkalns AL, Kushner LE, Stevens BA, Pinsky BA, Maldonado Y. Assessment of Sensitivity and Specificity of Patient-Collected Lower Nasal Specimens for Severe Acute Respiratory Syndrome Coronavirus 2Testing. JAMA Netw Open. 2020 Jun 1;3(6):e2012005. doi: 10.1001/jamanetworkopen.2020.12005. PMID 32530469
- [Background] Thirumurthy H, Masters SH, Mavedzenge SN, Maman S, Omanga E, Agot K. Promoting male partner HIV testing and safer sexual decision making through secondary distribution of self-tests by HIV-negative female sex workers and women receiving antenatal and post-partum care in Kenya: a cohort study. Lancet HIV. 2016 Jun;3(6):e266-74. doi: 10.1016/S2352-3018(16)00041-2. Epub 2016 Apr 8. PMID 27240789
- [Derived] Bien-Gund CH, Stephens-Shields AJ, Acri T, Dugosh K, Gross R. Provision of COVID-19 Self-Test Kits to Patients for Distribution to Social Contacts: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2513708. doi: 10.1001/jamanetworkopen.2025.13708. PMID 40465296

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Started | 395 | 397
Completed | 388 | 388
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Excluded due to administrative error | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution | Total
Number analyzed (Participants) | 388 | 388 | 776
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 352 | 352 | 704
  >=65 years | 36 | 36 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [32 to 58] | 44 [32 to 56] | 44 [32 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 individuals declined to answer.
  Participants
    number analyzed (Participants) | 387 | 387 | 774
    Female | 219 | 221 | 440
    Male | 168 | 166 | 334
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not all participants provided data or agreed to answer this question.
  Participants
    Hispanic or Latino | 53 | 59 | 112
    Not Hispanic or Latino | 322 | 318 | 640
    Unknown or Not Reported | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 230 | 249 | 479
  White | 88 | 69 | 157
  More than one race | 18 | 12 | 30
  Unknown or Not Reported | 37 | 40 | 77
Region of Enrollment [Number; unit: participants]
  United States | 388 | 388 | 776

OUTCOME MEASURES:

1. Primary Outcome: Network Contact Test Uptake
Description: The primary outcome is the proportion of study participants who distributed tests/referrals to least two network contacts who completed testing. This outcome will be measured by number of participants with at least 2 unique network contacts who completed a test linked to a study participant by week 8. The investigators will test for differences in the primary outcome between the two study arms.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 388 | 388
Participants | 5 | 2
Statistical Analysis 1: Comparison: Self-Test Kit Distribution vs Test Referral Distribution; Test type: Superiority; p = 0.45, Fisher Exact; Risk Difference (RD) = 0.0077, 95% CI 2-sided [-0.021 to 0.056]

2. Secondary Outcome: Network Contact Test Uptake, End of Study
Description: Test uptake among at least two network contacts. This outcome will be measured by the number of participants with at least two unique network contacts who completed a test linked to an index participant by end of study.
Time Frame: Through study completion, up to 30 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 388 | 388
Participants | 8 | 2
Statistical Analysis 1: Comparison: Self-Test Kit Distribution vs Test Referral Distribution; Test type: Superiority; p = 0.11, Fisher Exact; Risk Difference (RD) = 0.015, 95% CI 2-sided [-0.0004 to 0.03]

3. Secondary Outcome: Number of Contacts Tested at 8 Weeks
Description: Number of unique network contacts who completed a test linked to an index participant by week 8. Participants analyzed reflects the number of network contacts only who completed a test.
Time Frame: 8 weeks
Population: Note that each participant could have up to 5 network contacts, so the denominator = 5 times the number of index participants.
Measure: Count of Units; unit: Network contacts
Units Other Than Participants: Network contacts
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 388 | 388
Number analyzed (Network contacts) | 1940 | 1940
Network contacts | 23 | 13

4. Secondary Outcome: Number of Contacts Tested
Description: Number of unique network contacts who completed a test linked to an index participant by end of study.
Time Frame: Through study completion, up to 30 months
Population: as for outcome 3
Measure: Count of Units; unit: Network contacts
Units Other Than Participants: Network contacts
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 388 | 388
Number analyzed (Network contacts) | 1940 | 1940
Network contacts | 31 | 16

5. Secondary Outcome: Number of Participants With at Least One Network Contact Who Tested Positive for COVID-19 at 8 Weeks
Description: Number of participants with at least one network contact who tested positive for COVID-19 within 8 weeks of enrollment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 388 | 388
Participants | 3 | 0

6. Secondary Outcome: Number of Participants With at Least One Network Contact Who Tested Positive for COVID-19, End of Study
Description: Number of participants with at least one network contact who tested positive for COVID-19 by the end of study
Time Frame: Through study completion, up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
Number analyzed (Participants) | 388 | 388
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Subjects were considered enrolled in our study for 8 weeks. 8 weeks after enrollment, they completed a follow-up survey and were then considered to have completed the study. Note that network contacts could still continue testing for COVID-19 through study completion, up to 30 months.
Arm/Group | Self-Test Kit Distribution | Test Referral Distribution
All-Cause Mortality (participants affected / at risk) | 0/388 | 0/388
Serious Adverse Events (participants affected / at risk) | 0/388 | 0/388
Other Adverse Events (participants affected / at risk) | 0/388 | 0/388

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT04797858/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT04797858/ICF_001.pdf